CLINICAL TRIAL: NCT05053620
Title: Astigmatism Correction With Intrastromal Arcuate Incisions in Eyes Undergoing Cataract Surgery With Femtosecond Laser Using the Cassini Ambient With Iris Registration (ARCUATAS)
Acronym: ARCUATAS
Status: Completed | Type: Observational
Sponsor: OFTALVIST (Oftalmología Vistahermosa S.L) (Industry)
Collaborators: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARCUATAS
Record Dates: First submitted 2021-09-08; First posted 2021-09-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Single arm: All patients.
  Interventions: Device: Calculation of the arcuate intrasomal incisions

INTERVENTIONS:
Device: Calculation of the arcuate intrasomal incisions — All patients participating in the study will undergo femtosecond laser treatment for the correction of astigmatism through arcuate intrastromal incisions with the Catalys laser (Johnson & Johnson, USA, CE marked). The calculation of intrastromal arcuate incisions will be carried out using the following nomogram indicated on the laser: 9.0 mm optical zone and symmetrical incisions of 50 degrees for 0.50D, 55 degrees for 0.75D, 60 degrees for 1.00D and 65 degrees for 1.25D of corneal astigmatism. After the incisions, conventional cataract surgery will be performed using the Centurion phacoemulsifier equipment (Alcon, USA, with CE marking) in the ZCB00 monofocal intraocular lens (IOL) implant (Johnson & Johnson, USA, with CE marking). All patients will be treated according to standard clinical practice.

SUMMARY:
This is an observational, prospective follow-up post-marketing study of CE marked medical devices aimed at treating astigmatism in patients with cataracts. The main objective is to evaluate the response of the intrastromal arcuate incisions procedure for the correction of low corneal astigmatism with the Catalys femtosecond laser using the Cassini Ambient equipment with iris registration in cataract surgery.

DETAILED DESCRIPTION:
All patients participating in the study will undergo femtosecond laser treatment for the correction of astigmatism through arcuate intrastromal incisions with the Catalys laser (Johnson & Johnson, USA, CE marked). The calculation of intrastromal arcuate incisions will be carried out using the following nomogram indicated on the laser: 9.0 mm optical zone and symmetrical incisions of 50 degrees for 0.50D, 55 degrees for 0.75D, 60 degrees for 1.00D and 65 degrees for 1.25D of corneal astigmatism. After the incisions, conventional cataract surgery will be performed using the Centurion phacoemulsifier equipment (Alcon, USA, with CE marking) in the ZCB00 monofocal intraocular lens (IOL) implant (Johnson & Johnson, USA, with CE marking). All patients will be treated according to standard clinical practice.

A preoperative and postoperative evaluation will be carried out one month and four months after the intervention where the following tests will be performed: refraction, corneal topography with the Cassini Ambient equipment (Cassini Technologies, The Netherlands, with CE marking), measurement of visual acuity with and without correction, slit lamp examination and ocular biometry using the IOLMaster 700 non-contact optical biometer (Carl Zeiss, Germany, CE marked).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are going to undergo cataract surgery.
2. Low corneal astigmatism, between 0.50D and 1.25D.

Exclusion Criteria:

1. Previous corneal surgery.
2. Keratoconus.
3. Corneal scars
4. Pterygium
5. Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are already going to undergo conventional cataract surgery by phacoemulsification in which there is low corneal astigmatism (up to 1.25 D) and it is corrected by means of arcuate intrastromal incisions with femtosecond laser following routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Response to treatment | 4 months after the procedure
  Evaluation of the response to the procedure

SECONDARY OUTCOMES:
Evaluation of the visual acuity | 4 months after the procedure
  Evaluation of the visual acuity
Examination of the arcuate incisions | 4 months after the procedure
  Examination of the arcuate incisions using a slit amp

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Tañá Rivero, Doctor, Principal Investigator — OFTALVIST (Oftalmología Vistahermosa S.L)
Locations (1):
- OFTALVIST (Oftalmología Vistahermosa S.L.), Alicante, Spain

IPD SHARING:
Plan to Share IPD: No